CLINICAL TRIAL: NCT07128186
Title: The Application of an AI-driven Multimodal Predictive Model for Cognitive Impairment in Patients With Type 2 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yangyan, Principal Investigator, Tongji Hospital
Other Study IDs: TJ-IRB202503076
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Dysfunction
Keywords: mild cognitive impairment; type 2 diabetes mellitus; artificial intelligence-based multimodal cognitive screening system
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive Normal Group: Healthy control group without significant cognitive impairment in the study
  Interventions: Other: follow-up observation
- Mild Cognitive Impairment Group: An intermediate state with subjective or objective cognitive decline (e.g., memory, executive function) that does not meet the diagnostic criteria for dementia
  Interventions: Other: follow-up observation

INTERVENTIONS:
Other: follow-up observation — In this study, no additional interventions were administered to any enrolled participants; only 3-5 years of follow-up observation were conducted, with cognitive status data collected at both baseline and endpoint.

SUMMARY:
The objective of this observational study is to evaluate the accuracy and feasibility of an artificial intelligence-based multimodal cognitive screening system in early identification of diabetes-related mild cognitive impairment (MCI) among type 2 diabetes mellitus (T2DM) patients through a 3-5 year follow-up. It also aims to analyze the correlation between diabetic metabolic indicators (such as glycemic variability and HbA1c levels) and cognitive function changes, thereby determining the value of this intelligent screening system in early detection and intervention of cognitive impairment in T2DM patients, which constitutes the key focus of this research.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Diagnosed with type 2 diabetes mellitus (T2DM).
2. Aged 40-75 years, with self-reported or informant-reported memory complaints.
3. Cognitive assessment scores consistent with either:

   * Cognitive Normal (CN) or
   * Mild Cognitive Impairment (MCI).
4. Preserved ability to perform basic activities of daily living (ADLs).
5. Memory-specific deficits only (e.g., partial forgetfulness), with intact other cognitive domains (e.g., reasoning, judgment, attention, and executive function).

Exclusion Criteria:

1. Other types of diabetes (e.g., type 1 diabetes, gestational diabetes).
2. Education level <6 years.
3. Metabolic disorders that may affect cognition, including:

   * Acute carbohydrate metabolism events within 3 months (e.g., severe hypoglycemia, diabetic ketoacidosis, hyperglycemic hyperosmolar state).
   * Hypothyroidism or other endocrine disorders.
4. Neurological/psychiatric conditions that may impair cognition:

   * History of head trauma, depression, anxiety, delirium, severe pulmonary/renal disease, heart failure, or malignancy.
5. Substance abuse (past 2 years), including nicotine/alcohol dependence.
6. Recent medication use (within 1 month):

   * Anti-Parkinsonian drugs, antiepileptics, sedatives/hypnotics.
7. Cognitive-enhancing drugs (e.g., donepezil, memantine).
8. Inability to complete AI screening or follow-up due to:

   * Speech/hearing/visual impairments or other disabilities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll 5,000 eligible participants from 20 participating centers across Hubei Province for a 3- to 5-year longitudinal follow-up, with strict adherence to the predefined inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Early Identification Accuracy of the AI System | From enrollment to the end of follow-up for 3-5 years
  Sensitivity, specificity, and area under the ROC curve (AUC) of the AI system in detecting Mild Cognitive Impairment (MCI), compared with traditional scales (MMSE/MoCA).
Cognitive Deterioration Rate | From enrollment to the end of follow-up for 3-5 years
  Conversion rates from:Cognitively Normal (CN) → MCI; MCI → Alzheimer's Disease (AD)

SECONDARY OUTCOMES:
Association Between Diabetic Metabolic Indicators and Cognitive Decline | From enrollment to the end of follow-up for 3-5 years
  Correlation of glucose variability (e.g., MAGE) and glycated hemoglobin (HbA1c) with changes in cognitive scores.
Predictive Value of Multimodal Data | From enrollment to the end of follow-up for 3-5 years
  Predictive efficacy of voice features, facial expressions, drawing trajectories, and other biomarkers in forecasting cognitive deterioration

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Minda Hospital Affiliated to Hubei Minzu University, Enshi, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - Huangshi Central Hospital, Huangshi, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Sinopharm Dongfeng General Hospital, Shiyan, Hubei
  - Suizhou Central Hospital, Suizhou, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - China Resources & WISCO General Hospital, Wuhan, Hubei
  - Hubei Provincial Hospital of Integrated Chinese & Western Medicine, Wuhan, Hubei
  - Tianyou Hospital Affiliated to Wuhan University of Science and Technology, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan Fifth Hospital, Wuhan, Hubei
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangyang First People's Hospital, Xiangyang, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - Xiantao First People's Hospital, Xiantao, Hubei
  - Xiaogan Central Hospital, Xiaogan, Hubei
  - Renhe Hospital Affiliated to China Three Gorges University, Yichang, Hubei
  - Sinopharm Gezhouba Central Hospital, Yichang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei